CLINICAL TRIAL: NCT01974622
Title: Indocyanine Green Angiography-Guided Photodynamic Therapy for Treatment of Retinal Capillary Abnormalities.
Brief Title: ICG-Guided Photodynamic Therapy for Treatment of Retinal Capillary Abnormalities: A Pilot Study
Acronym: ICGguidedPDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG- guided PDT Study
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Retinal Vascular Disorders
MeSH Terms: interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Visudyne (Experimental): Visudyne half fluence- 1 treatment with the possibility of a second treatment.
  Interventions: Drug: Visudyne

INTERVENTIONS:
Drug: Visudyne — Half fluence verteporfin
  Other Names: Verteporfin

SUMMARY:
The purpose of this research is to use an approved drug(Visudyne) for neovascular age-related macular degeneration, which is essentially choroidal neovascularization for permeability and vascular proliferation for the retinal circulation, to treat another permeable abnormality - retinal capillary abnormalities - located eccentric to the central portion of the macula or in the foveal region.

DETAILED DESCRIPTION:
The study will include 30 patients who were diagnosed with retinal capillary abnormalities and include 2 follow-up visits at 6 and 12 months post-procedure to determine if the treatment has been effective in treating their disorder. It is anticipated that approximately half of the patients will require an additional treatment. Patients will be enrolled from our patient population and be 50 years of age and older, male or female. Pregnant women or women of normal child bearing age will be excluded since there are no adequate and well-controlled studies on the use of photodynamic therapy in pregnant women. Any retinal vascular abnormality that has a standard of care method of treatment will also be excluded from the study population.

ELIGIBILITY:
Inclusion Criteria:• Individuals that are 50 years of age and older.

* Patients with retinal capilary abnormalities/vascular diseases such as macular telangiectasia type I and type II, retinal arteriolar macroanurysms, and retinal angiomous proliferation (RAP).
* Patients with diabetic retinopathy and branch retinal vein occlusions
* Other patients who are non-responders to approved treatment methods

Exclusion Criteria:

* Patients whose diseases have approved methods of treatment.
* Pregnant women or women of normal child bearing age.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Improvement and/or stabilization of disease. | 1-2 years
  The drug, approved for are-related macular degeneration should also prove effective for other permeable conditions, such as retinal capillary/vascular abnormalities that lead to macular edemas such as macular telangiectasia type I and type II, retinal arteriolar macroanurysms, and retinal angiomatous proliferation (RAP), which is a variant of neovascular age-related macular degeneration. These diseases currently have no available approved alternative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, M.D., Principal Investigator — Northshore LIJ/MEETH
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

REFERENCES:
- [Background] Yannuzzi LA, Slakter JS, Gross NE, Spaide RF, Costa DL, Huang SJ, Klancnik JM Jr, Aizman A. Indocyanine green angiography-guided photodynamic therapy for treatment of chronic central serous chorioretinopathy: a pilot study. 2003. Retina. 2012 Feb;32 Suppl 1:288-98. doi: 10.1097/iae.0b013e31823f99a9. PMID 22451952